CLINICAL TRIAL: NCT01889225
Title: Obesity and Mortality
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Allison, Phd, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: R01-DK076771-Aim1A; R01DK076771 (NIH)
Record Dates: First submitted 2013-06-20; First posted 2013-06-28 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (19):
- Multiple Risk Factor Intervention Trial - Usual Group
- Multiple Risk Factor Intervention Trial - Referred Group
- Framingham Heart study
- Framingham Offspring cohort
- Atherosclerosis Risk In Communities
- Charleston Heart study
- Cardiovascular Health study
- Rancho Bernardo study
- Nurses' Health I study
- Panel Study Income Dynamics
- MRFIT Referred Care
- HDFP Referral Care
- Alameda County Health and Ways of Living Study
- Nurses' Health II study
- Tecumseh County Health study
- EPESE-East Boston: Established Populations for Epidemiologic Studies of the Elderly-East Boston
- EPESE-Duke: Established Populations for Epidemiologic Studies of the Elderly-Duke
- EPESE-Iowa: Established Populations for Epidemiologic Studies of the Elderly-Iowa
- EPESE-New Haven: Established Populations for Epidemiologic Studies of the Elderly-New Haven

SUMMARY:
Previous analyses of the National Health and Nutrition Examination Survey have suggested that the mortality rate associated with obesity has decreased over calendar time in the U.S. population, potentially due to improvements in the medical care of obesity and its associated diseases. The primary aim of this project is to evaluate whether this reduction in the detrimental association of obesity with mortality rate over calendar time is supported by other data from U.S. prospective studies.

ELIGIBILITY:
Inclusion Criteria:

* U.S. based studies with at least 1500 subjects
* At least 5 years of mortality follow-up
* BMI measured or self-reported available at 2 or more separate calendar time
* Subjects varied in age at baseline

Exclusion Criteria:

* Any study that does not meet the inclusion criteria was excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: U.S. based prospective cohorts of adults
Sampling Method: Non-Probability Sample
Enrollment: 311982 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Years of Life Lost Associated with Standard BMI categories Over Calendar Time | Between 1960 and 2000 (up to 40 years)

SECONDARY OUTCOMES:
Change in Adjusted Hazard Ratio Over Calendar Time for Standard BMI Categories | Between 1960 and 2000 (up to 40 years)

CONTACTS AND LOCATIONS:
Overall Officials: David B Allison, Ph.D., Principal Investigator — University of Alabama at Birmingham